CLINICAL TRIAL: NCT01363180
Title: Stress-induced Drinking in Emerging Adults: the Role of Trauma History
Acronym: ARC5
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: P50AA010761-16 (NIH)
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Trauma; Posttraumatic Stress Disorder
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control
  Interventions: Behavioral: Trier Social Stress Test (TSST); Other: No stress condition
- Trauma-exposed without PTSD
  Interventions: Behavioral: Trier Social Stress Test (TSST); Other: No stress condition
- Trauma-exposed with PTSD
  Interventions: Behavioral: Trier Social Stress Test (TSST); Other: No stress condition

INTERVENTIONS:
Behavioral: Trier Social Stress Test (TSST) — The TSST is a standardized psychological stress challenge where a participant performs a speech and mental math task in front of 3 unfamiliar individuals, in order to evoke an HPA axis stress response in a laboratory setting.
Other: No stress condition

SUMMARY:
This project is the first to use a clinical laboratory method in emerging adults to test the hypothesis that a trauma history with or without concommitant posttraumatic stress disorder (PTSD) alters response to a stressor and promotes drinking compared to normal controls. The study will be the first to explore whether trauma-exposed (TE) and PTSD groups differ on these outcomes. It will also examine the relationship between stress reactivity and subsequent stress-induced drinking in these samples. The goal of this program is to better understand the relationship between stress and factors related to the development and maintenance of alcohol problems in early adults, so that ultimately, better treatments may be developed that reduce the incidence and severity of alcohol related problems.

DETAILED DESCRIPTION:
This study will be conducted with a 3 x 2 between subjects design. The between groups factors are (1) trauma group (3 levels: Control, Trauma Exposed with, and without PTSD) and (2) exposure to stress (2 levels: yes and no). To decrease intra-group variability, trauma type will be limited to interpersonal trauma. Potential participants will be screened over the phone. Those meeting basic eligibility criteria will complete an assessment at the MUSC Institute of Psychiatry, and those meeting final eligibility criteria will be scheduled for the laboratory session to be completed at the Clinical and Translational Research Center (CTRC).

Half of each trauma history group will receive the Trier Social Stress Test (TSST); the other half will receive a no-stress control condition. Baseline and post-stress objective and subjective measures of stress reactivity will be collected. Following the stress task, all participants will be given a priming dose and subsequently presented with an alcohol taste test. The primary analyses will examine the effect of trauma group membership on response to stress and subsequent voluntary drinking. Based on power analyses using preliminary data from similar samples, a sample size of 240 participants (40 per cell) is required.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-30 years old.
* Must drink alcohol on at least 4 days in the past month.
* Must drink beer (thought not necessarily exclusively)
* Must be able to read and provide informed consent.
* Trauma history group criteria:
* To be eligible for Control group, participants must not have a history of Criteria A traumatic event(s), as defined by the DSM-IV.
* To be eligible for the Trauma-Exposed group (TE), participants must have a history of a Criteria A traumatic event that involves interpersonal violence, but not meet DSM-IV criteria for PTSD (current or lifetime)as defined by the MINI, and a PCL score 20 or below.
* To be eligible for the PTSD group, participants must have a history of exposure to a Criteria A traumatic event that involves interpersonal violence, currently meet criteria for PTSD (defined by DSM-IV) and a PCL score of 30 or above.

Exclusion Criteria:

* Currently taking psychoactive medication, antihistamines, or medication that alters HPA axis functioning.
* Severe obesity (BMI > 40)
* Current alcohol dependence.
* Current abuse or dependence on illicit substances (with the exceptions of caffeine and nicotine)
* Smokers who cannot abstain from smoking for at least 4 hours.
* Current major depression.
* Current or lifetime psychosis.
* Any medical condition that impacts HPA axis functioning.
* Any blood clotting disorder.
* Pregnant or nursing women, or women who suspect that may be pregnant.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 21-30 year olds
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla K Danielson, Ph.D., Principal Investigator — Medical University of South Carolina; Suzanne Thomas, Ph.D., Study Director — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- See also: MUSC Clinical Trials Registry — http://www.scresearch.org